CLINICAL TRIAL: NCT05997134
Title: Assessment of Three Regimens of Ketamine Infusion in Complex Regional Pain Syndrome: Randomized Prospective Comparative Study
Brief Title: Three Regimens of Ketamine Infusion in Complex Regional Pain Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aml Magdy Abo Elsafa, resident of anesthesiology, surgical intensive care and pain medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MS44/1/23
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Ketamine Infusion; Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Ketamine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): patients will receive ketamine parenteral infusion (0.35 mg/kg/h or maximum 24mg/h) at post anesthetic care unit(PACU) over 6 hours for 3days
  Interventions: Drug: Ketamine
- Group B (Experimental): patients will receive ketamine parenteral infusion (0.35 mg/kg/h or maximum 24mg/h ) at post anesthetic care unit(PACU) over 6 hours for 5 days .
  Interventions: Drug: Ketamine
- Group C (Experimental): patients will receive ketamine parenteral infusion (0.35 mg/kg/h or maximum 24mg/h ) at post anesthetic care unit(PACU) over 6 hours for 7 days
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — patients will receive ketamine parenteral infusion (0.35 mg/kg/h or maximum 24mg/h) at post anesthetic care unit(PACU) over 6 hours for 3days .
  Arms: Group A
Drug: Ketamine — patients will receive ketamine parenteral infusion (0.35 mg/kg/h or maximum 24mg/h ) at post anesthetic care unit(PACU) over 6 hours for 5 days
  Arms: Group B
Drug: Ketamine — patients will receive ketamine parenteral infusion (0.35 mg/kg/h or maximum 24mg/h ) at post anesthetic care unit(PACU) over 6 hours for 7 days
  Arms: Group C

SUMMARY:
To evaluate the efficacy of three regimens of sub anesthetic dose of ketamine infusion in relieving chronic refractory pain in patients with complex regional pain syndrome

DETAILED DESCRIPTION:
Ketamine N-methyl-D-aspartate (NMDA) receptor blocker that has recently been studied for its analgesic effect is a phencyclidine or phenyl cyclohexyl piperidine (PCP) derivative that initially became commercially available for human use in 1970 as a rapid-acting intravenous (IV) anesthetic. It is currently classified by the Food and Drug Administration (FDA) as an anesthetic induction agent in doses ranging from 1 to 4.5 mg/kg.

Ketamine has proven to be a desirable drug, despite of its induction dissociative effects and abuse potential. It is favorable due to its short half-life and lack of clinically significant respiratory depression. In addition to its anesthetic effects, ketamine has analgesic, anti-inflammatory, and antidepressant activities.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 21 years old of both sexes with American Standards Association I ,II.
* Patients diagnosed as ( CRPS) based on Budapest criteria
* The average daily pain intensity required on (NRS) is 7 or more for at least 3 months despite of standard therapy which includes: (pharmacologic therapy as non steroidal anti- inflammatory drugs (NSAIDs), antiepileptic (AEDs), antidepressants), as well as physical therapy and psychiatric care

Exclusion Criteria:

* patients refusal
* Patients with unstable psychological or psychiatric conditions, including : untreated bipolar disorder, post-traumatic stress disorder, major depression , severe personality disorder and psychotic illness.
* Patients have recently undergone major interventional pain procedures, such as nerve blocks or implantable therapies within 3 months of enrollment.
* Patients with known drug dependency or substance use disorder specifically related to ketamine or other psycho-stimulant drugs.
* Patients with previous severe reactions, contraindication or allergy to ketamine.
* Patients with cardiovascular disease (hypertension, arrhythmia), hepatic, renal or other organ impairment.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
degree of chronic pain reduction | up to 3 months post infusion
  using Brief Pain Inventory short form (BPI-SF) questionnaire. It is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10 point scale.

SECONDARY OUTCOMES:
Reduction of the degree of chronic pain score | up to 3 months post infusion
  Numerical rating scales (NRS) is an 11-point scale for patient self-reporting of pain. It is based solely on the ability to perform activities of daily living (ADLs) with 0 being "no pain" and 10 being "the worst pain imaginable"
Side effects | up to 3 months post infusion
  Headache, Nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-garbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol, CSR
Time Frame: after the end of study for one year
Access Criteria: The data will be available upon a reasonable request from the corresponding author